CLINICAL TRIAL: NCT03996356
Title: Clozapine Induced Weight Gain: A Pharmacogenetic Study
Brief Title: Clozapine Induced Weight Gain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CT/688/000000/16
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Weight Gain; Antipsychotic Agents; Pharmacogenetics
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 blood samples to be taken at 0 and 6 months (2x EDTA plasma/whole blood, 2x serum).
  Biochemical markers and status of 2 common single nucleotide polymorphisms will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No study intervention - observational study — This is an observational study where the comparative groups will be determined by the genetic variants (SNPs) of subjects and not an intervention, per se.

SUMMARY:
Clozapine is prescribed to patients with psychosis in whom other treatments have not worked. Research has shown, however, that clozapine may be associated with weight gain and abnormal blood sugar levels in some patients. There is strong evidence to suggest that genetic variation between individuals plays an important role in the development of these side effects in response to the medication. Our research aims to evaluate the effects of two genes and the blood level of clozapine on side-effects such as weight changes and blood sugar levels in patients receiving clozapine treatment. From out-patient clinics in Cwm Taf UHB, the investigators aim to recruit 160 patients who are taking clozapine; collect information/ measurements from recruits relating to size/ weight/ BMI, risk of diabetes and blood samples to measure markers of blood sugar, fat/lipids, clozapine and its breakdown products, blood cells and variants of two specific genes. From this information the investigators will be particularly interested to understand if there is any association between the variation in these two genes with weight gain or changes in blood sugar, in patients taking clozapine.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Taking/compliant with clozapine antipsychotic medications.
* Patients meeting the ICD-10 criteria for a diagnosis of schizophrenia, schizoaffective or borderline personality disorders.

Exclusion Criteria:

* History of current alcohol/illicit substance dependency.
* Unable/ unsuitable to complete the study protocol e.g. acutely ill, suicidal or aggressive patients.
* Unable to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on clozapine treatment
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Body-mass index (BMI) | 12 months
  BMI will be calculated by weight (kg)/ height^2 (m^2).
Leptin gene promoter region single nucleotide polymorphisms (SNPs) (rs7799039) | 12 months
  SNPs will be determined by polymerase chain reaction followed by restriction fragment length polymorphism analysis to determine (c.-2548G or c.-2548A) .
Serotonin 5-HT 2C receptor gene single nucleotide polymorphisms (SNPs) (rs3813929) | 12 months
  SNPs will be determined by polymerase chain reaction followed by restriction fragment length polymorphism analysis to determine (c.-759C or c.-759T) .

SECONDARY OUTCOMES:
Blood haemoglobin A1c concentration | 6 months
  Haemoglobin A1c concentrations will be determined by ion-exchange HPLC (G8, Tosoh, Amsterdam, Netherlands)
Waist:hip ratio | 12 months
  Waist:hip ratio will be calculated by waist circumference (cm)/hips circumference (cm)
Lipid profile | 12 months
  Serum lipid profiles will include total cholesterol, HDL cholesterol, LDL cholesterol and triglyceride. These will be measured by enzymatic colorimetric methods on cobas-Roche analysers (Roche, Burges Hill, UK) except LDL cholesterol, which will be calculated using the Friedewald equation ([LDL cholesterol] = [Total cholesterol] - ([Triglyceride] / 2.2) - [HDL cholesterol]
Clozapine side effects assessment by Clinical Global Impression (CGI) scale | 12 months
  Clinical Global Impression (CGI) scale is a validated tool to assess clozapine side effects (Ref: Guy W, editor. ECDEU Assessment Manual for Psychopharmacology. 1976. Rockville,MD, U.S. Department of Health, Education, and Welfare)
Clozapine:nor clozapine ratio | 12 months
  Clozapine:nor clozapine ratio is calculated by clozapine (ug/L)/ nor clozapine (ug/L) both measured by high-performance liquid chromatography with diode-array detection.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Tennant, PhD, Principal Investigator — Cwm Taf Morgannwg UHB
Locations (1):
- Cwm Taf University Health Board, Merthyr Tydfil, Wales, United Kingdom

REFERENCES:
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Baptista T, Kin NM, Beaulieu S, de Baptista EA. Obesity and related metabolic abnormalities during antipsychotic drug administration: mechanisms, management and research perspectives. Pharmacopsychiatry. 2002 Nov;35(6):205-19. doi: 10.1055/s-2002-36391. PMID 12518268
- [Background] Basile VS, Masellis M, McIntyre RS, Meltzer HY, Lieberman JA, Kennedy JL. Genetic dissection of atypical antipsychotic-induced weight gain: novel preliminary data on the pharmacogenetic puzzle. J Clin Psychiatry. 2001;62 Suppl 23:45-66. PMID 11603885
- [Background] Couchman L, Morgan PE, Spencer EP, Flanagan RJ. Plasma clozapine, norclozapine, and the clozapine:norclozapine ratio in relation to prescribed dose and other factors: data from a therapeutic drug monitoring service, 1993-2007. Ther Drug Monit. 2010 Aug;32(4):438-47. doi: 10.1097/FTD.0b013e3181dad1fb. PMID 20463634
- [Background] Mammes O, Betoulle D, Aubert R, Herbeth B, Siest G, Fumeron F. Association of the G-2548A polymorphism in the 5' region of the LEP gene with overweight. Ann Hum Genet. 2000 Sep;64(Pt 5):391-4. doi: 10.1017/s0003480000008277. PMID 11281277
- [Background] Mantzoros CS. The role of leptin in human obesity and disease: a review of current evidence. Ann Intern Med. 1999 Apr 20;130(8):671-80. doi: 10.7326/0003-4819-130-8-199904200-00014. PMID 10215564
- [Background] Ohlson LO, Larsson B, Svardsudd K, Welin L, Eriksson H, Wilhelmsen L, Bjorntorp P, Tibblin G. The influence of body fat distribution on the incidence of diabetes mellitus. 13.5 years of follow-up of the participants in the study of men born in 1913. Diabetes. 1985 Oct;34(10):1055-8. doi: 10.2337/diab.34.10.1055. PMID 4043554
- [Background] Reynolds GP, Zhang ZJ, Zhang XB. Association of antipsychotic drug-induced weight gain with a 5-HT2C receptor gene polymorphism. Lancet. 2002 Jun 15;359(9323):2086-7. doi: 10.1016/S0140-6736(02)08913-4. PMID 12086765
- [Background] Reynolds GP, Zhang Z, Zhang X. Polymorphism of the promoter region of the serotonin 5-HT(2C) receptor gene and clozapine-induced weight gain. Am J Psychiatry. 2003 Apr;160(4):677-9. doi: 10.1176/appi.ajp.160.4.677. PMID 12668355